CLINICAL TRIAL: NCT01848392
Title: Extra Pulmonary Determinants of Physical Activity in Adults With Cystic Fibrosis.
Brief Title: Extrapulmonary Effects of Cystic Fibrosis on Physical Activity of Adult Patients.
Acronym: MUCO-DAP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: 2011 - A00819 - 32
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Adults; Physical activity
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- physical activity CF cohort: adult patients with CF at time of their yearly assessment at Cochin adult CF centre

SUMMARY:
Physical activity seems to be a prognostic factor for quality of life and survival in patients with cystic fibrosis (CF). Whereas their exercise capacity has been assessed through medical examination, their daily physical activity has been little studied. Activity monitors have measured physical activity only in a few studies which considered mainly respiratory status and more recently bone mineral density and body composition. Determinants of physical activity in patients with CF remain largely unknown.

The objective of this study is to measure daily physical activity with activity monitors in adult patients with CF and to investigate the determinants of physical activity, with a focus on extra-respiratory factors (nutritional status, diabetes, bone mineralization, anxiety and/or depression, cardiac impairment).

Seventy adult patients with CF, regularly cared at the Cochin adult CF centre, will be recruited in a stable period during their annual review. During this assessment, laboratory tests will be carried out (especially parameters for nutritional status), as well as measurement of body composition and bone mineral density, respiratory function tests and a 6 minute walk test, and echocardiography. Patients will wear for 7 consecutive days a multi-sensor armband SenseWear on the arm, to assess the intensity of physical activity in metabolic equivalents (METS) and steps per day. Finally, patients will complete three self-administered questionnaires: Quality of Life (CFQ14 +), hospital anxiety depression scale and physical activity.

After a descriptive analysis of the study cohort, we will study qualitative and quantitative criteria related to physical activity (assessed quantitatively by the number of steps/day or metabolic equivalents).

Linear regression models will then be developed to assess the independent factors associated with physical activity, adjusting for different variables of interest related to patients demographic, behavioral, clinical (respiratory and non-respiratory ) and biological parameters. Conversely, the "predictive" independent aspect of physical activity will be studied according to respiratory function, nutritional status and quality of life.

DETAILED DESCRIPTION:
Ambulatory adult CF patients are recruited at time of their yearly evaluation.

Phenotypic patients' characteristics Age, gender, CFTR genotype, pancreatic status (presence or absence of exocrine pancreatic insufficiency), number of IV antibiotic courses and number of hospitalization over the previous year, are reported.

Physical activity measurement Physical activity is measured over 7 consecutive days using a multisensor armband (SenseWear Pro Armband; BodyMedia, Inc.,Pittsburgh, PA) that is worn on the upper right arm over the triceps muscle. It incorporates a biaxial accelerometer that records steps per day, and physiologic indicators of energy expenditure that enable the investigator to determine the physical activity level.

Evaluation of respiratory function and cardiovascular status Patients will perform a respiratory function test to evaluate FVC and FEV1 and six minutes walk test. Arterial blood gases will be done at the beginning and at the end of walk and the walking distance will be indicated in meters.

Echocardiography will be performed to look for left or right cardiac dysfunction and measure systolic pulmonary artery pressure. N-terminal pro-B-type natriuretic peptide (NT-pro-BNP) will be used as a systemic biomarker of heart failure.

Bone mineral density (BMD) and body composition They are measured by X-ray absorptiometry (DEXA) on the lumbar spine, femur and whole body, and measurement of lean and fat mass (Lunar Prodigy).

Nutritional evaluation Weight and height are measured and body mass index (BMI) is calculated. As part of the annual dietary assessment, there will be an evaluation of the amount of ingested nitrogen.

Blood will be drawn to measure: albumin, prealbumin, vitamin E, vitamin A and vitamin 25(OH)D3, HbA1c. C-reactive protein and fibrinogen will be measured as indicators of inflammation.

Urinalysis will measure: creatinine, nitrogen and 3-methylhistidine. Oral glucose tolerance test will be performed (fasting blood glucose and blood glucose 2 hours after ingesting 75 g of glucose) in pancreatic insufficient patients with unknown diabetes.

Self-administered questionnaires

Patients will answer 3 questionnaires:

1. quality of life CFQ14+ questionnaire
2. hospital anxiety depression (HAD) scale validated in French
3. Baecke physical activity questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients with CF (positive sweat test or 2 disease causing CFTR mutations)
* Aged 18 or older
* Regularly cared at Cochin adult CF centre
* In clinical stable status

Exclusion Criteria:

* Pulmonary exacerbation in the 4 previous weeks
* IV antibiotic course for pulmonary exacerbation in the 2 previous weeks
* Pregnancy in female patients
* Patient with history of lung transplantation
* Patient on a waiting list for lung transplantation
* Treatment of diabetes initiated for less than 3 months
* Enteral nutrition initiated for less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with CF cared at Cochin adult CF centre, Paris
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-02-21 (Actual); Primary Completion 2014-07-30 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
Steps per day | Day 7
  The armband indicates the mean number of steps per day over a 7-day period
Physical activity level | Day 7
  The investigators determine the physical activity level by dividing total daily energy expenditure by whole-night sleeping energy expenditure

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hubert, MD, Principal Investigator — Université Paris-Centre, AP-HP
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Troosters T, Langer D, Vrijsen B, Segers J, Wouters K, Janssens W, Gosselink R, Decramer M, Dupont L. Skeletal muscle weakness, exercise tolerance and physical activity in adults with cystic fibrosis. Eur Respir J. 2009 Jan;33(1):99-106. doi: 10.1183/09031936.00091607. Epub 2008 Aug 20. PMID 18715878
- [Background] Tejero Garcia S, Giraldez Sanchez MA, Cejudo P, Quintana Gallego E, Dapena J, Garcia Jimenez R, Cano Luis P, Gomez de Terreros I. Bone health, daily physical activity, and exercise tolerance in patients with cystic fibrosis. Chest. 2011 Aug;140(2):475-481. doi: 10.1378/chest.10-1508. Epub 2011 Feb 3. PMID 21292759
- [Background] Watz H, Waschki B, Boehme C, Claussen M, Meyer T, Magnussen H. Extrapulmonary effects of chronic obstructive pulmonary disease on physical activity: a cross-sectional study. Am J Respir Crit Care Med. 2008 Apr 1;177(7):743-51. doi: 10.1164/rccm.200707-1011OC. Epub 2007 Nov 29. PMID 18048807